CLINICAL TRIAL: NCT06557343
Title: Single-Cell Sequencing Analysis of Radiation Pneumonitis Signals In Patients Treated For Cancer With Radiotherapy
Acronym: SPITFIRE
Status: Recruiting | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 339413
Record Dates: First submitted 2024-06-03; First posted 2024-08-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Radiation Pneumonitis
Keywords: radiation pneumonitis; cancer; single cell sequencing
MeSH Terms: conditions — Radiation Pneumonitis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoscopy sample (deep bronchial brushing) producing cellular fluid sample for processing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bronchoscopy under ELFMAN: Clinical bronchoscopy performed under ELMAN study
  Interventions: Diagnostic Test: Single Cell Sequencing

INTERVENTIONS:
Diagnostic Test: Single Cell Sequencing — Sequencing of all viable single cells present in deep bronchial brushings using transcriptomics to identify what cells are present and what they are doing.

SUMMARY:
Patients with signs of radiation induced lung inflammation, who are referred for a clinical bronchoscopy for investigation, will have a sample sent for single cell sequencing. This is a novel technique which allows for identification of which cells are present and what they are doing. This hopes to better understand radiation pneumonitis, a dose-limiting toxicity in cancer treatment which can be highly morbid and even fatal.

DETAILED DESCRIPTION:
Lung cancer is the third most common cancer in the UK with around 48,500 people diagnosed with the condition each year. Unfortunately, despite significant progress in treatment options and their delivery, improvements in survival remain elusive. Radiotherapy (RT) is a cornerstone of both radical and palliative treatment in non-small cell lung cancer (NSCLC). Radiation pneumonitis (RP) is the key dose-limiting constraint and a morbid, potentially even life-threatening, toxicity associated with RT to the thorax. Newer combinations of chemo-radiotherapy and adjuvant immunotherapy demonstrate improved survival but are associated with higher risk of RP.

Current management of RP is very limited consisting of supportive measures and steroids; the latter of which are often ineffective and come with their own risks. The typical triad of symptoms (exertional dyspnoea, a non-productive cough and hypoxia) can be directly fatal for some whilst for others represent a devastating and permanent decline in their lung function and quality of life. Although modest understanding of the patient and treatment related risk factors for RP development have been identified the underlying mechanisms remain poorly understood and has been challenging to investigate. A cascade of inflammatory changes with hypoxia lead to endovascular damage, cytokine release and ultimately endothelial cell death and irreversible fibrosis. Single-cell RNA sequencing (scRNA-seq) is a relatively novel technique that allows access to an understanding of this process. It can allow the identification of what genetics, cell types and functional heterogeneity are up/down-regulated in association with irradiated lung tissue in humans.

It is known that Stereotactic-Ablative Radiotherapy (SABR) is a well-tolerated highly conformal form of RT. It has been safely delivered to patients before radical surgery without significant toxicity or increase in complication rate. If a targetable mechanism behind this condition could be identified it has the potential to change the landscape of lung cancer RT management and in doing so save lives.

A literature search revealed no investigation like this has been conducted in humans. A Chinese study has been done in murine models and demonstrated several signals which, if demonstrated in humans, could be of interest. SPITFIRE proposes to obtain inflamed lung tissue from patients who have developed pneumonitis following radiation for their lung cancer to find these answers.

1.2 RATIONALE FOR STUDY Both patients who have potentially been cured of their lung cancer and those being treated to alleviate symptoms in their last months-to-years of life are diagnosed with RP. Potentially treatable disease can be refused due to an unacceptable combination of risk factors for developing RP. Hospitalisation for RP is common and yet often frustratingly unhelpful. RP is a major contributor to patient morbidity, mortality and healthcare cost. Although clearly a constant concern in lung cancer any radiation delivered through the chest (including oesophageal, breast and pulmonary metastatic RT) carries a risk of RP.

Pulmonary fibrosis treatment is starting to improve with novel agents such as Nintedanib and Pirfenidone demonstrating some promise. There is likely, though yet unproven, crossover between the molecular and genetic processes involved in these conditions. Should a better understanding of the mechanisms behind RP reveal a targetable signal, and subsequent treatment, it has the potential to completely change not only the management of this toxicity but that of thoracic malignancies.

Obtaining tissue from human lung affected by RP is a challenge. These patients are often too unstable to safely proceed with such intervention. There is, however, a population of patients who have clinical and radiological features diagnostic of the condition but maintain oxygen saturations (SpO2) adequate to proceed to bronchoscopy. Some of these patients will be referred for a bronchoscopy to exclude super-added infection. As part of this process they may be enrolled in the ELFMAN (Edinburgh Lung Fibrosis Molecular Endotyping) Study - to better characterise suspected inflammatory and fibrotic interstitial lung disease, as it may have shared molecular pathways to interstitial pneumonias including idiopathic pulmonary fibrosis (IPF). Standard bronchoscopy may not reach the effect area of lung but deep bronchial brushings obtains a good cellular yield which should be adequate for scRNA-seq whilst minimising risk to the patient. This study proposes to utilise a brushing from these patients to process using a novel laboratory technique to help identify the cellular processes that may be involved in radiation pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient has received thoracic radiotherapy and has clinical or radiological features in fitting with a diagnosis of Radiation Pneumonitis (onset one to four months post-RT with breathlessness, especially exertional, cough, chest discomfort, which is persistent over weeks, a chest x-ray [CXR] may demonstrate patchy or widespread opacification although can be normal.)
* Must be ambulant, oxygen independent with SpO2 >92% on air and haemodynamically stable to be considered safe for a bronchoscopy.
* Willing to undergo and likely able to tolerate bronchoscopy, ie. Can lie flat without compromising ventilation, and able to consent to the ELFMAN Protocol and SPITFIRE trial.

Exclusion Criteria:

* Contraindication to bronchoscopy, ie. Previously not tolerated, unable to lie flat, Sp02 <92% on air
* Patient requires admission or oxygen dependant
* Test positive for Covid-19 within the preceding six weeks to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the above eligibility criteria who demonstrate clinical/radiological diagnosis of radiation pneumonitis
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful creation of dataset | within a month of sample collection, a year to recruit five patients
  If deep bronchial brushings generates sufficient viable cells for processing via single-cell sequencing this will generate a dataset of cellular activity for each of these five patients. The only way to know if this technique - ie. the use of deep bronchial brushings combined with single-cell sequencing, is to run the test on the samples and therefore successful generation of the dataset is proof of feasibility of the method. There may be further use for this dataset (ie. secondary outcome below) but primarily this process will prove feasibility simply by generating data. This is not a health outcome, simply demonstration of a viable sample using a novel combination of sampling and laboratory test.

SECONDARY OUTCOMES:
Signals in pneumonitis | 3-6 months
  Comparison with normal lung dataset (publicly available) to potentially identify radiation pneumonitis signals that may be targetable via drug therapy or worth expanding to a larger trial to explore.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Centre for Information Research, University of Edinburgh, Edinburgh
  - Henderson Lab, Edinburgh
  - Edinburgh Cancer Centre, Edinburgh

IPD SHARING:
Plan to Share IPD: No
Linked anonymized data only